CLINICAL TRIAL: NCT06677853
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II/III Clinical Study to Evaluate the Efficacy and Safety of Timolol Maleate Gel in the Treatment of Proliferating Superficial Infantile Hemangioma
Brief Title: Timolol Maleate Gel for the Treatment of Infantile Hemangioma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Auson Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN001C002; ASN001C002 (Registry Identifier: China Drug Trials)
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Infantile Hemangioma
Keywords: superficial; proliferating; Infantile Hemangioma; Timolol Maleate
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Intervention Model Description: It was a multicenter, randomized, double-blind, placebo-controlled Phase II/III clinical study to evaluate the efficacy and the safety of TM gel in the treatment of superficial IH in the proliferative phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group1-Timolol Maleate Gel + Placebo (Experimental): 56 patients will be randomized to group 1.
  Interventions: Drug: Timolol Maleate Gel+Placebo
- Group 2-Timolol Maleate Gel (Experimental): 56 patients will be randomized to group 2.
  Interventions: Drug: Timolol Maleate Gel
- Group 3-Placebo (Placebo Comparator): 56 patients will be randomized to group 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Timolol Maleate Gel+Placebo — Subjects were applied with the 0.5% timolol maleate gel at the affected area twice a day, and with the placebo once a day for 24 weeks.
  Arms: Group1-Timolol Maleate Gel + Placebo
Drug: Timolol Maleate Gel — Subjects were applied with the 0.5% timolol maleate gel at the affected area 3 times a day for 24 weeks.
  Arms: Group 2-Timolol Maleate Gel
Drug: Placebo — Subjects were applied with placebo at the affected area 3 times a day for 24 weeks.
  Arms: Group 3-Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of timolol maleate (TM) gel in subjects with superficial infantile hemangioma (IH) in the proliferative phase. The main question it aims to answer is:

• The primary endpoint (success or failure) assessment was a centralized and independent qualitative assessment based on blinded comparison on B-ultrasonography results and photographs of IH at W24 from baseline.

Researchers will compare TM gel to a placebo (a look-alike substance that contains no drug) to see if TM gel works to treat IH.

Participants will:

* Take the study drug 3 times daily (once in the morning, noon, and evening, respectively) for 24 weeks.
* The family members of patients are instructed to bring the patients to the clinic for regular follow-up visits at Week 4 (W4), Week 12 (W12), and Week 24 (W24) of the treatment period.
* Keep a diary of concomitant medications and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants at the age of 35 ~ 150 days;
2. Infant subjects with definitive diagnosis of superficial hemangioma requiring treatment based on medical history, clinical manifestations, and imaging examination (B-ultrasonography, CT or MRI) results;
3. Infant subjects with single hemangioma lesion;
4. Infant subjects with the maximum hemangioma diameter being ≥ 1 cm but ≤ 10 cm;
5. Infant subject with CEA ≥ Grade 2; The guardians of the infant subject understood the study contents and risks of study treatment, signed the informed consent form (ICF), and were willing to cooperate with the study conduct.

Exclusion Criteria:

1. Infant subjects who were known to be allergic to or had history of severe allergy to timolol maleate or other β-receptor blockers;
2. Infant subjects who had previously been treated with systemic, intralesional or topical corticosteroids, vincristine, α-interferon, imiquimod, propranolol, or other β-receptor blockers;
3. Infant subjects breastfed by mother who was treated with β-receptor blockers, systemic (oral, intravenous or intramuscular) corticosteroids, vincristine or α-interferon while breastfeeding;
4. Infant subjects who born more than 2 months premature and younger than 60 days old;
5. Infant subjects who had previously been treated for hemangioma (including surgery, hormonal drugs, laser therapy, etc.);
6. Infant subjects with more than one type of hemangioma requiring treatment;
7. Infant subjects with other skin diseases on the hemangioma surface and surrounding skin areas, such as eczema, infantile eczema, etc.
8. Infant subjects who had atrioventricular block ≥ second-degree, bradycardia (heart rate < 100 bpm), sinoatrial syndrome, cardiogenic shock, or other congenital cardiac disorders;
9. Infant subjects who were suffering from respiratory disorders such as bronchial asthma, bronchospasm and pneumonia;
10. Infant subjects who were suffering from central nervous system disorders, or had symptoms of increased intracranial pressure, or had other underlying diseases that might cause or aggravate infantile hemangioma;
11. Infant subjects who had systolic blood pressure < 50 mmHg or diastolic blood pressure < 30 mmHg;
12. Infant subjects who received any other investigational drug within 4 weeks prior to screening; Infant subjects with other conditions not suitable for enrollment at the discretion of the investigator.

Ages: 35 Days to 150 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Success rate of cure of IH after 24-week treatment. | 24 weeks
  Treatment success is defined as complete or almost complete resolution of the patient's IH at W24 compared with baseline.
  At the time of centralized independent assessment.

SECONDARY OUTCOMES:
Changes in the hemangioma volume | baseline, week 4, 12 and 24
  Changes in the hemangioma volume from baseline after treatment for 4, 12 and 24 weeks, adopting the estimation formula of IH volume: V = 0.07×(the average of the hemangioma's longest length and width)^3.
Changes in hemangioma color | baseline, weeks 4, 12 and 24
  Change in the color of hemangioma after 4, 12, and 24 weeks of treatment, which is assessed by the CEA (Clinician Erythema Assessment) criteria.The color intensity (e.g., no signs of erythema;slight redness;defined redness;marked redness;fiery redness.) of the IH is assessed on a 5 point scale.
Complete/almost complete regression rates of IH from baseline after 4 and 12-week treatment. | baseline, weeks 4 and 12
  At the time of centralized independent assessment.
Complete/almost complete resolution rate of IH at each post-baseline visit (Weeks 4, 12, and 24) from baseline. | baseline, Weeks 4, 12, and 24
  On-site qualitative assessment by the investigator of efficacy.
Evolution of IH at each post-baseline visit(Weeks 4, 12, and 24) from baseline. | baseline, Weeks 4, 12 and 24
  Classified into 5 categories: completely/almost completely resolved, improved, stable, aggravated, and not assessable.
  On-site qualitative assessment by the investigator of efficacy.
Changes in IH at each post-baseline visit(Weeks 4, 12, and 24) compared to the previous visit. | Baseline, Weeks 4, 12, and 24
  Classified into 5 categories: complete/almost complete regression, relief, stabilization, exacerbation, and unable to determine.
  On-site qualitative assessment by the investigator of efficacy.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital, Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanxi, Taiyuan, Shanxi
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Kunming Children's Hospital, Kunming, Yunan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No